CLINICAL TRIAL: NCT03591406
Title: An Open-label, Randomised Controlled Multi-centre Study to Assess the Impact of Ferric Carboxymaltose in Correcting Iron Deficiency Anaemia Compared With Venofer® (Iron Sucrose) in Chinese Subjects
Brief Title: To Assess the Impact of Ferric Carboxymaltose Compared With Iron Sucrose in Chinese Subjects on Correcting Iron Deficiency Anaemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vifor (International) Inc. (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIT-IRON-2011-004
Record Dates: First submitted 2018-06-22; First posted 2018-07-19 (Actual); Results first posted 2020-05-18 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; Ferric Oxide, Saccharated

STUDY DESIGN:
Intervention Model Description: Open-label, parallel design, randomised controlled multi-centre trial in Chinese subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferric carboxymaltose (FCM) (Experimental): Subjects treated with FCM given by IV injection or drip infusion
  Interventions: Drug: Ferric carboxymaltose
- Iron sucrose (IS) (Active Comparator): Subjects treated with IS given by IV injection or drip infusion
  Interventions: Drug: Iron sucrose

INTERVENTIONS:
Drug: Ferric carboxymaltose — Dosage Form: Injection, Sterile FCM solution as a 5% w/v iron solution in water for injection Strength: 10 mL vials containing 500 mg iron per vial Dosage: 500mg/week or 1000mg/week (based on subject BW and Hb value at screening) Route of administration: IV injection (undiluted solution) or drip infusion (500 mg iron diluted in 100 mL 0.9% w/v physiological saline or 1,000 mg iron diluted in 250 mL 0.9% w/v physiological saline) Dosing schedules: baseline (Day 1) and, if required, at Day 8 and Day 15.
  Other Names: FCM
  Arms: Ferric carboxymaltose (FCM)
Drug: Iron sucrose — Dosage Form: Sterile solution for injection containing 2% w/v iron Strength: 5 mL ampoules containing 100 mg iron per ampoule Dosage: single doses of IS of 200mg iron based on the formula of Ganzoni: Cumulative iron deficit [mg] = BW [kg] x (target Hb- actual Hb) [g/dL] x 2.4 + 500 mg, up to 11 IS injections will be given Route of administration: IV injection or drip infusion Dosing schedules: three times a week, with an initial dose at baseline and will receive iron, as per approved label, until the subject has received the calculated iron dose.
  Other Names: IS; Venofer™
  Arms: Iron sucrose (IS)

SUMMARY:
The primary objective is to demonstrate the efficacy of ferric carboxymaltose (FCM) given in a simple dosing regimen in correcting iron deficiency anaemia (IDA), by demonstrating non-inferiority to treatment with the currently approved intravenous (IV) iron therapy of iron sucrose (IS, Venofer™) in the Chinese population. The secondary objectives are to assess the safety of FCM compared to IS in the Chinese population and to evaluate the effect of FCM compared to IS on relevant laboratory parameters (haematology, chemistry, iron parameters) in the Chinese population.

DETAILED DESCRIPTION:
This is an open-label, randomised controlled study to assess the impact of FCM in correcting iron deficiency anaemia compared with Venofer™ (IS).

All subjects, after providing written informed consent and meeting the eligibility assessments, will receive a first dose of IV iron as either FCM or IS. A total of approximately 368 subjects (184 per group) will be enrolled. All subjects will have iron deficiency anaemia as measured by haemoglobin (Hb), serum ferritin and transferrin saturation (TSAT) at screening.

Ferric carboxymaltose will be administered as either a diluted infusion or undiluted injection (at Investigator discretion) and IS will be administered as a slow intravenous injection at a rate of 1 ml undiluted solution per minute (with each single injection of 200 mg iron) or by drip infusion. Note, for subjects randomised to receive IS dosing visits are required three times a week to achieve total iron repletion dosing as calculated using the Ganzoni formula.

For subjects randomised to FCM, the total iron requirements will be calculated at screening based on the screening Hb and subject weight. Dosing will be at baseline and, if required, at day 8 and day 15. All subjects will attend study visits at screening, baseline and thereafter at Weeks 2, 4 and 6. All subjects will attend an end of study visit (at Week 8 - or earlier if discontinued prematurely).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Hb <11 g/dL (females) or Hb <12 g/dL (males) at the screening visit
* Serum ferritin <100 ng/mL for subjects with underlying inflammatory disease (e.g., inflammatory bowel disease (IBD), chronic kidney disease (CKD) or chronic heart failure (CHF), as determined by high sensitive C-reactive protein [hsCRP] levels above the normal range) otherwise ≤14 ng/mL in subjects with no apparent underlying inflammatory disease (as determined by hsCRP levels within normal range) at the screening visit
* Transferrin Saturation (TSAT) <16% (any subject) at the screening visit
* Microcytic, hypochromic anaemia defined as: a) Mean corpuscular Hb concentration (MCHC) <32%; b) Mean corpuscular volume (MCV) < 80 fL; c)Mean corpuscular Hb (MCH) <27 pg
* Subjects with the ability to understand the requirements of the study and abide by the study restrictions, and who agree to return for the required assessments
* Before any study-specific procedure is conducted, the appropriate written informed consent must be obtained

Exclusion Criteria:

* Subject has known hypersensitivity to any of the products to be administered during dosing
* Any history of iron storage diseases such as haemochromatosis
* Any history or clinical findings of iron utilisation disorders such as sideroachrestic anaemia
* Known haemoglobinopathy (e.g. thalassaemia)
* Any history or clinical findings of anaemia associated with: a) Haematuria b) Vitamin B12 or folic acid deficiency that requires treatment (subjects can be included after deficiency is corrected)
* Any allergic predispositions, i.e. any history of asthma or atopic allergy. This includes drug allergies.
* Planned surgery with anticipated blood loss (defined as Hb drop >2 g/dL) in the 3 months post randomisation
* Subject has known malignancy (with or without current treatment), except basal cell or squamous cell carcinoma of the skin or cervical intra-epithelial neoplasia
* Haemodialysis (current or planned within the next 3 months)
* History of IV iron therapy, erythropoiesis stimulating agent (ESA) therapy and/or blood transfusion in previous 4 weeks prior to screening, and oral iron or oral iron-containing products including Chinese herbal medicines (>75mg iron/day) in the 7 days prior to screening
* Body weight <35 kg
* Chronic liver disease and/or screening alanine transaminase (ALT) or aspartate transaminase (AST) above 3 times the upper limit of the normal range
* Known human immunodeficiency virus infection, acquired immunodeficiency syndrome, tuberculosis
* Known active hepatitis B or C or other active infection (acute or chronic)
* Subject currently is enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study(ies), or subject is receiving other investigational agent(s)
* Subject is pregnant or is breast feeding
* Female subject of childbearing potential not using adequate contraceptive methods during the study and for up to 1 month after the last dose of the study medication. Adequate contraceptive methods are defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intra-uterine devices, sexual abstinence or vasectomised partner. Non-childbearing potential includes being surgically sterilised at least 6 months prior to the study or post-menopausal, defined as amenorrhoea for at least 12 months
* Male subjects planning to father a child within 7 days from the last study drug administration.
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures and/or other reason(s) that render subject not appropriate for study participation in the opinion of the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, Principal Investigator — The First Affiliated Hospital, Zhejiang University; Zhihua Ran, Principal Investigator — Renji Hospital Shanghai Jiaotong Uniersity School of Medicine
Locations (1):
- The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang, China

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects who provided signed and dated informed consent were screened within 7 days prior to initial treatment administration.
Groups:
- Ferric Carboxymaltose (FCM): Participants treated with FCM given by IV injection or drip infusion
  Dosage Form: Injection, Sterile FCM solution as a 5% w/v iron solution in water for injection
  Strength: 10 mL vials containing 500 mg iron per vial
  Dosage: 500mg/week or 1000mg/week (based on subject Body Weight (BW) and Hb value at screening)
  Route of administration: IV injection (undiluted solution) or drip infusion (500 mg iron diluted in 100 mL 0.9% w/v physiological saline or 1,000 mg iron diluted in 250 mL 0.9% w/v physiological saline)
  Dosing schedules: baseline (Day 1) and, if required, at Day 8 and Day 15.
- Iron Sucrose (IS): Participants treated with IS given by IV injection or drip infusion
  Dosage Form: Sterile solution for injection containing 2% w/v iron
  Strength: 5 mL ampoules containing 100 mg iron per ampoule
  Dosage: single doses of IS of 200mg iron based on the formula of Ganzoni: Cumulative iron deficit [mg] = BW [kg] x (target Hb- actual Hb) [g/dL] x 2.4 + 500 mg, up to 11 IS injections will be given
  Route of administration: IV injection or drip infusion
  Dosing schedules: three times a week, with an initial dose at baseline and will receive iron, as per approved label, until the subject has received the calculated iron dose.
Period: Overall Study
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (IS)
Started | 188 | 183
Completed | 181 | 174
Not Completed | 7 | 9
Not completed — Adverse Event | 5 | 3
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 0 | 5

BASELINE CHARACTERISTICS:
Population: Demography and baseline characteristics for the Safety Set (SS) are provided. The SS was defined as all randomised subjects who received at least 1 dose of study medication.
Groups:
- Ferric Carboxymaltose (FCM): Participants treated with FCM given by IV injection or drip infusion
  Dosage Form: Injection, Sterile FCM solution as a 5% w/v iron solution in water for injection
  Strength: 10 mL vials containing 500 mg iron per vial
  Dosage: 500mg/week or 1000mg/week (based on subject BW and Hb value at screening)
  Route of administration: IV injection (undiluted solution) or drip infusion (500 mg iron diluted in 100 mL 0.9% w/v physiological saline or 1,000 mg iron diluted in 250 mL 0.9% w/v physiological saline)
  Dosing schedules: baseline (Day 1) and, if required, at Day 8 and Day 15.
- Total: Total of all reporting groups
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (IS) | Total
Number analyzed (Participants) | 187 | 180 | 367
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (9.85) | 38.9 (8.70) | 39.4 (9.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 169 | 342
  Male | 14 | 11 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 187 | 180 | 367
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 187 | 180 | 367
Haemoglobin [Mean (Standard Deviation); unit: g/dl] | 7.74 (1.491) | 8.06 (1.453) | 7.90 (1.479)
Serum ferritin [Mean (Standard Deviation); unit: ng/ml] | 4.47 (2.145) | 4.93 (6.095) | 4.70 (4.534)
Transferrin saturation (TSAT) [Mean (Standard Deviation); unit: %] | 4.82 (1.898) | 4.92 (2.912) | 4.87 (2.446)
High-sensitivity C-reactive protein (hsCRP) [Mean (Standard Deviation); unit: mg/l] | 1.026 (2.1432) | 1.567 (5.9817) | 1.291 (4.4617)

OUTCOME MEASURES:

1. Primary Outcome: Participants Achieving an Increase in Hb of at Least 2 g/dL at Any Time up to Week 8
Description: Haemoglobin (Hb)
Time Frame: From baseline at any time up to Week 8
Population: Per Protocol Set: participants who were randomised, received at least 1 dose of study treatment, had at least 1 baseline and post-baseline value (Hb, ferritin, TSAT), had a study drug compliance between 80% and 120% and had no major protocol violations
Measure: Count of Participants; unit: Participants
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (IS)
Number analyzed (Participants) | 177 | 178
Participants | 176 | 175
Statistical Analysis 1: Comparison: Ferric Carboxymaltose (FCM) vs Iron Sucrose (IS); Test type: Non-Inferiority — Pre-defined non-inferiority margin of -15%; Difference in proportions = 1.12, 95% CI 2-sided [-2.15 to 4.71] — 2-sided 95% Confidence Interval (CI) was computed using the Wilson score method with continuity correction described by Newcombe

2. Secondary Outcome: Participants Achieving an Increase in Hb of at Least 2 g/dL From Baseline to Weeks 2, 4, 6 and 8
Description: Haemoglobin (Hb)
Time Frame: From Baseline to weeks 2, 4, 6 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (IS)
Number analyzed (Participants) | 177 | 178
Participants
  Week 2: number analyzed (Participants) | 176 | 177
  Week 2 | 150 | 129
  Week 4: number analyzed (Participants) | 172 | 173
  Week 4 | 164 | 167
  Week 6: number analyzed (Participants) | 173 | 172
  Week 6 | 169 | 168
  Week 8: number analyzed (Participants) | 175 | 173
  Week 8 | 173 | 171

3. Secondary Outcome: Change in Hb From Baseline to Weeks 2, 4, 6, and 8
Description: Haemoglobin (Hb)
Time Frame: From Baseline to weeks 2, 4, 6 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (IS)
Number analyzed (Participants) | 177 | 178
g/dL
  Week 2: number analyzed (Participants) | 176 | 177
  Week 2 | 3.01 (1.135) | 2.53 (1.016)
  Week 4: number analyzed (Participants) | 172 | 173
  Week 4 | 4.46 (1.502) | 4.08 (1.217)
  Week 6: number analyzed (Participants) | 173 | 172
  Week 6 | 4.96 (1.435) | 4.61 (1.422)
  Week 8: number analyzed (Participants) | 175 | 173
  Week 8 | 5.09 (1.504) | 4.87 (1.525)

4. Secondary Outcome: Participants With Iron Deficiency Correction Over Time by Treatment
Description: Iron deficiency correction: TSAT >= 16% and serum ferritin >=100ng/mL (for subjects with underlying inflammatory disease) or >14ng/mL (for subjects with no apparent underlying inflammatory disease).
Time Frame: From Baseline to Weeks 2, 4, 6 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (IS)
Number analyzed (Participants) | 177 | 178
Participants
  Week 2: number analyzed (Participants) | 176 | 170
  Week 2 | 173 | 135
  Week 4: number analyzed (Participants) | 171 | 173
  Week 4 | 165 | 168
  Week 6: number analyzed (Participants) | 174 | 172
  Week 6 | 161 | 163
  Week 8: number analyzed (Participants) | 175 | 173
  Week 8 | 162 | 154

5. Secondary Outcome: Change in TSAT From Baseline to Weeks 2, 4, 6 and 8
Description: Transferrin saturation (TSAT)
Time Frame: From Baseline to weeks 2, 4, 6 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of TSAT
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (IS)
Number analyzed (Participants) | 177 | 178
Percentage of TSAT
  Week 2 | 30.16 (11.741) | 25.03 (19.474)
  Week 4 | 28.00 (8.528) | 25.30 (8.453)
  Week 6 | 25.50 (9.097) | 23.33 (7.868)
  Week 8 | 25.32 (10.793) | 20.82 (7.618)

6. Secondary Outcome: Change in Serum Ferritin From Baseline to Weeks 2, 4, 6 and 8
Time Frame: From Baseline to Weeks 2, 4, 6 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (IS)
Number analyzed (Participants) | 177 | 178
ng/ml
  Week 2: number analyzed (Participants) | 176 | 177
  Week 2 | 759.72 (331.118) | 385.51 (145.647)
  Week 4: number analyzed (Participants) | 171 | 173
  Week 4 | 379.31 (195.415) | 280.58 (148.913)
  Week 6: number analyzed (Participants) | 174 | 172
  Week 6 | 255.71 (152.582) | 184.93 (100.677)
  Week 8: number analyzed (Participants) | 175 | 173
  Week 8 | 202.09 (148.382) | 145.56 (89.890)

7. Secondary Outcome: Change in Serum Iron From Baseline to Weeks 2, 4, 6 and 8
Time Frame: From Baseline to weeks 2, 4, 6 and 8
Population: Safety Set: all randomised participants who have received at least 1 dose of study medication. The participants in this group were analysed based on the treatment they received.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (IS)
Number analyzed (Participants) | 187 | 180
umol/L
  Week 2: number analyzed (Participants) | 185 | 179
  Week 2 | 15.53 (7.075) | 16.23 (14.512)
  Week 4: number analyzed (Participants) | 178 | 173
  Week 4 | 12.31 (4.209) | 12.39 (4.724)
  Week 6: number analyzed (Participants) | 180 | 172
  Week 6 | 10.77 (4.318) | 11.27 (4.160)
  Week 8: number analyzed (Participants) | 181 | 175
  Week 8 | 10.77 (4.871) | 10.09 (4.152)

8. Secondary Outcome: Participants With Any Treatment Emergent Adverse Event (TEAE)
Description: Please note that in this section we are presenting just the overview of the adverse events experienced by the trial participant, in particular, the number of participants with at least one TEAE until end of the trial.
  Please refer to the detailed tables included on the Adverse Event Module for specifics
Time Frame: From Baseline to the End of the study (week 8)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (IS)
Number analyzed (Participants) | 187 | 180
Participants | 124 | 101

9. Secondary Outcome: Blood Pressure at Baseline and Weeks 2, 4, 6 and 8
Description: Diastolic Blood pressure
Time Frame: Baseline and weeks 2, 4, 6 and 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (IS)
Number analyzed (Participants) | 187 | 180
mmHg
  Baseline | 69.8 (7.91) | 71.9 (8.85)
  Week 2: number analyzed (Participants) | 185 | 179
  Week 2 | 71.0 (8.33) | 72.6 (8.79)
  Week 4: number analyzed (Participants) | 179 | 173
  Week 4 | 72.1 (7.60) | 73.8 (9.57)
  Week 6: number analyzed (Participants) | 180 | 173
  Week 6 | 71.6 (8.18) | 74.3 (9.24)
  Week 8: number analyzed (Participants) | 181 | 175
  Week 8 | 72.4 (8.09) | 74.1 (9.77)

10. Secondary Outcome: Body Weight at Baseline and Week 8
Time Frame: Baseline and week 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (IS)
Number analyzed (Participants) | 187 | 180
kg
  Baseline | 59.76 (9.384) | 60.40 (9.354)
  Week 8: number analyzed (Participants) | 181 | 175
  Week 8 | 59.73 (9.316) | 60.64 (9.372)

11. Secondary Outcome: Heart Rate at Baseline and Weeks 2, 4, 6 and 8
Time Frame: Baseline and weeks 2, 4, 6 and 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (IS)
Number analyzed (Participants) | 187 | 180
beats/min
  Baseline | 81.4 (8.85) | 82.2 (9.94)
  Week 2: number analyzed (Participants) | 185 | 179
  Week 2 | 76.3 (9.80) | 76.5 (8.83)
  Week 4: number analyzed (Participants) | 179 | 173
  Week 4 | 75.5 (10.71) | 76.6 (10.79)
  Week 6: number analyzed (Participants) | 180 | 173
  Week 6 | 76.0 (8.98) | 77.2 (10.04)
  Week 8: number analyzed (Participants) | 181 | 175
  Week 8 | 75.8 (10.33) | 77.5 (10.94)

12. Secondary Outcome: Body Temperature at Baseline and Weeks 2, 4, 6 and 8
Time Frame: Baseline and weeks 2, 4, 6 and 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ºC
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (IS)
Number analyzed (Participants) | 187 | 180
ºC
  Baseline | 36.94 (0.292) | 36.45 (0.325)
  Week 2: number analyzed (Participants) | 185 | 179
  Week 2 | 36.48 (0.269) | 36.44 (0.288)
  Week 4: number analyzed (Participants) | 179 | 173
  Week 4 | 36.49 (0.269) | 36.40 (0.268)
  Week 6: number analyzed (Participants) | 180 | 173
  Week 6 | 36.47 (0.259) | 36.41 (0.260)
  Week 8: number analyzed (Participants) | 181 | 175
  Week 8 | 36.48 (0.269) | 36.46 (0.257)

ADVERSE EVENTS:
Time Frame: From Baseline until the End of the Study (8 weeks)
Description: All AEs either observed by the Investigator/collaborators, or reported by the subject spontaneously, or in response to a direct question, were noted in the AE section of the case report form/source document. In order to avoid bias in eliciting AEs, subjects were asked a non-leading question, such as "How are you feeling?" A non-leading question was used as well for changes in their health or concomitant medication usage since their last visit. This information was collected at all study visits.
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Sucrose (IS)
All-Cause Mortality (participants affected / at risk) | 0/187 | 0/180
Serious Adverse Events (participants affected / at risk) | 10/187 | 7/180
Other Adverse Events (participants affected / at risk) | 124/187 | 92/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferric Carboxymaltose (FCM) (N=187) | Iron Sucrose (IS) (N=180)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic adhesions (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferric Carboxymaltose (FCM) (N=187) | Iron Sucrose (IS) (N=180)
Urine phosphorus decreased (Investigations) | 14 (18) | 14 (16)
Blood phosphorus decreased (Investigations) | 13 (13) | 1 (1)
Alanine aminotransferase increased (Investigations) | 11 (14) | 5 (6)
White blood cells urine positive (Investigations) | 7 (7) | 8 (8)
Aspartate aminotransferase increased (Investigations) | 7 (7) | 4 (4)
Gamma-glutamyl transferase increased (Investigations) | 6 (6) | 6 (6)
Hepatic enzyme increased (Investigations) | 6 (7) | 3 (3)
Red blood cells urine positive (Investigations) | 4 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 15 (17) | 13 (13)
Urinary tract infection (Infections and infestations) | 6 (6) | 7 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 19 (20) | 5 (5)
Nausea (Gastrointestinal disorders) | 5 (6) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 2 (2) | 4 (4)
Pyrexia (General disorders) | 12 (12) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 13 (16) | 9 (12)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 2 (2) | 6 (6)
Headache (Nervous system disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT03591406/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/06/NCT03591406/SAP_001.pdf